CLINICAL TRIAL: NCT03547297
Title: INSIGHT-AHP: A Study to Characterize the Prevalence of Acute Hepatic Porphyria (AHP) in Patients With Clinical Presentation and History Consistent With AHP
Status: Terminated | Type: Observational
Why Stopped: Sponsor elected not to continue with study
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-AS1-NT-002
Record Dates: First submitted 2018-05-18; First posted 2018-06-06 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Acute Hepatic Porphyria; Hepatic Porphyrias; Acute Intermittent Porphyria (AIP); Hereditary Coproporphyria (HCP); Variegate Porphyria (VP); ALA Dehydratase Deficient Porphyria (ADP); Porphyria Acute
Keywords: Acute Hepatic Porphyria; Hepatic Porphyrias; Acute Intermittent Porphyria (AIP); Hereditary Coproporphyria (HCP); Variegate Porphyria (VP); ALA Dehydratase Deficient Porphyria (ADP); Porphyria Acute
MeSH Terms: conditions — Coproporphyria, Hereditary; Porphyrias, Hepatic; Porphyria, Acute Intermittent; Porphyria, Variegate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will use specific diagnostic tests on a group of patients who are experiencing symptoms typical of acute hepatic porphyria (AHP) to determine how many have the condition, and to potentially help improve the diagnostic process for patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age
* Recurrent and severe episodes of abdominal pain that last for at least 24 hours
* At least 1 episode of severe abdominal pain that required an urgent healthcare visit in the past 12 months
* Other symptoms related to AHP that your doctor will discuss with you
* Willing and able to comply with protocol required assessments and provide written informed consent

Exclusion Criteria:

* Known diagnosis of AHP
* Alternative explanation for abdominal pain with clinical response to treatment specific for alternative diagnosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female participants age ≥ 16 years who present with symptoms consistent with Acute Hepatic Porphyria such as recurrent and severe episodes of abdominal pain.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with current or past clinically symptomatic AHP with urinary aminolevulinic acid (ALA) or porphobilinogen (PBG) values above the upper limit of normal (ULN) | 12 months

SECONDARY OUTCOMES:
Proportion of participants with AHPs that contain likely pathogenic mutation(s) in the presence of urinary ALA or PBG values above the ULN | 12 months
Proportion of patients with pathogenic mutation(s) in the presence of urinary ALA and PBG values above the ULN | 12 months
Proportion of patients with variants of unknown significance in the presence of urinary ALA and PBG values above the ULN | 12 months
Proportion of patients with negative genetic tests in the presence of urinary ALA or PBG values above the ULN | 12 months
Correlation of biochemical and genetic test results with severity of disease measured by symptom frequency and severity in the participant questionnaire | 12 months
Correlation of biochemical and genetic test results with severity of disease measured by healthcare utilization in the participant questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Quinn Dinh, MD, Study Director — Alnylam Pharmaceuticals
Locations (12):
- United States (12):
  - Clinical Trial Site, Pasadena, California
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Margate, Florida
  - Clinical Trial Site, Ames, Iowa
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Manhasset, New York
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Pottsville, Pennsylvania
  - Clinical Trial Site, Knoxville, Tennessee
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided